CLINICAL TRIAL: NCT06879444
Title: "Investigation of 'Core' Stabilization Strength and Pelvic Floor Functions in Individuals with Primary Sjogren: a Controlled Study"
Brief Title: "Core Stabilization Strenght and Pelvic Floor Functions in Primary Sjogren's"
Status: Enrolling by invitation | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Begüm AKAR, Principal investigator, Pamukkale University
Other Study IDs: Pamukkale U
Record Dates: First submitted 2025-02-24; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Sjogren Syndrome; Healthy Volunteers
Keywords: pelvic floor; core stabilization; Sjogren syndrome
MeSH Terms: conditions — Sjogren's Syndrome | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- control group: The control group will consist of healthy volunteers.
  Interventions: Other: Core Muscle testing and patient reported outcome measures
- Sjogren syndrome: The Sjogren syndrome group will consist of patients aged between 18-65 who apply to the Rheumatology Department of Pamukkale University and meet the inclusion criteria.
  Interventions: Other: Core Muscle testing and patient reported outcome measures

INTERVENTIONS:
Other: Core Muscle testing and patient reported outcome measures — These are the situation evaluation parameters. It presents the data of the participants at the time of evaluation.

SUMMARY:
This study aims to explain the comparison of core stabilization strength and pelvic floor functions between individuals diagnosed with Sjogren syndrome and a healthy control group.

(Sjogren syndrome group n=27; control group n=27)

ELIGIBILITY:
Inclusion Criteria:

Sjogren syndrome group:

* Diagnosed by a rheumatologist
* Being 18 years of age or older,
* Agreeing to participate in the study

Control group:

-Being 18 years of age or older,

Exclusion Criteria:

Sjogren syndrome group and control group:

* Presence of neurological disease
* Presence of any orthopedic problem that would affect functionality
* Presence of a history of orthopedic surgery

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Sjogren syndrome group and control group
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2025-04-05 (Estimated); Study Completion 2025-06-05 (Estimated)

PRIMARY OUTCOMES:
Pelvic Floor Distress Inventory-20 (PTDE-20) | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  There are 20 questions in total on the scale. The best score that can be obtained from the entire survey is "0" and the worst score is "300".
Sexual Life Quality Scale- Women (CYKÖ-K) | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  The maximum score that can be obtained from the scale with this system is 108.
Incontinence Impact Questionnaire (IIQ-7) (IES) | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  Consists of 7 items. Maximum score is 100.
The McGill trunk muscle endurance test | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  The McGill trunk muscle endurance test is a test group that includes all trunk flexor, extensor and lateral muscle endurance tests.

SECONDARY OUTCOMES:
Health assessment questionnaire (HAQ) | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  This questionnaire consists of 20 questions and 8 subheadings, each answer ranging from 0 to 3 points.
Cognitive Exercise Therapy Approach (BETY) | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  This scale has 30 items. The scale is scored with a 5-point Likert system.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale Üniversitesi, Denizli, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Akar B, Kabul EG, Calik BB, Bozcuk S, Cobankara V. Investigation of Core Stabilization Strength and Pelvic Floor Functions in Patients with Primary Sjogren's Syndrome: A Case-Control Study. Int Urogynecol J. 2026 Jan 15. doi: 10.1007/s00192-025-06467-6. Online ahead of print. PMID 41538013